CLINICAL TRIAL: NCT02387684
Title: Efficay of Extended Peginterferon Alpha 2a(PEG-IFN a-2a) Treatment in HBeAg Negative Chronic Hepatitis B Patients
Brief Title: Efficay of Extended Peginterferon Alpha 2a Treatment in HBeAg Negative Chronic Hepatitis B Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, liver diseases center, Beijing Ditan Hospital
Other Study IDs: DTXY007
Record Dates: First submitted 2015-03-01; First posted 2015-03-13 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B; interferon; peginterferon; HBsAg loss
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The most important method to slow down and stop the liver disease progression in patients with chronic hepatitis B is antiviral therapy, by which to achieve maintaining viral response during treatment or obtain sustained viral response after treatment. The aim of the therapy with interferon is make patients obtain immune control to HBV defined as sustained viral response after treatment, however, most patients can't get this target after 48 weeks of interferon treatment, and some patients need extended treatment in clinical practice to enhance the rate of sustained viral response or HBsAg loss occurred during treatment. In this cohort study, the efficacy of extended therapy of interferon in HBeAg negative chronic hepatitis B patients will be evaluated.

DETAILED DESCRIPTION:
In this cohort study, the HBeAg negative chronic hepatitis B patients would be treated with peginterferon alpha 2a(PEG-IFN a-2a) for 96 week and followed 24 weeks after treatment. Serum HBV DNA load, HBsAg/anti-HBs level, HBeAg/anti-HBe will be tested at enrollment and every 3 months during treatment and follow period. Parameters of liver and kidney function, and liver ultrasound examination will be tested with intervals 1-3 months. The efficacies were evaluated by the rate of HBsAg loss during treatment and the rate of sustained viral response after treatment and follow up.

ELIGIBILITY:
Inclusion Criteria:

* HBeAg negative chronic hepatitis B patients

Exclusion Criteria:

* Active consumption of alcohol and/or drugs
* Co-infection with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus
* History of autoimmune hepatitis
* Psychiatric disease
* Evidence of neoplastic diseases of the liver

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Population in this cohort study was composed of HBeAg negative chronic hepatitis B patients defined as HBsAg positive, HBeAg negative,and detectable HBV DNA load with ALT level ≥41 U/L for more than 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
rate of sustained viral response | 120 weeks
  Sutained viral response was defined as serum HBV DNA undetectable at the end of treatment and the end of 24 weeks follow up.

SECONDARY OUTCOMES:
rate of HBsAg loss | 96 weeks
  HBsAg loss was defined as HBsAg level lower than 0.05 IU/ml.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan hospital,Capital Medical University, Beijing, Beijing Municipality, China